CLINICAL TRIAL: NCT00272233
Title: Effects of Sleep Loss on Endothelial Function and Cytokine Levels in Internal Medicine Residents
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Other Study IDs: HIC26414; NIH NHLBI K24 04024
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2006-01

CONDITIONS: Sleep Deprivation
Keywords: Inflammation Mediators [D23.469]; Cardiovascular Physiologic Phenomena [G09.330.553]
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Work requirements for medical trainees result in substantial sleep loss. Sleep loss has been associated with increased levels of certain inflammatory hormones that could have negative impact on blood vessel function. The purpose of this study is to determine the effects of sleep loss on blood hormone levels and blood vessel function in medical trainees.

DETAILED DESCRIPTION:
Context: Sleep loss is associated with increased blood levels of interleukin-6 (IL-6) and C-reactive protein (CRP). Medical residents are often deprived of normal sleep during extended work shifts, but the effects of work-related sleep loss on biomarkers of vascular inflammation and function are unknown.

Objective: We sought to test the hypothesis that sleep loss during extended work shifts during medical training is associated with increased circulating levels of pro-inflammatory biomarkers and evidence of vascular dysfunction.

Design: Outcome measures were assessed after extended 30-hour work shifts and non-extended 6-hour work shifts in a single-blind, randomized crossover design.

Setting: University hospital medical intensive care unit

Patients or Other Participants: Twenty-two healthy medical residents were studied during a medical intensive care unit rotation.

Main Outcome Measure(s): Sleep related cytokines (interleukin-6 and tumor necrosis factor), serum markers of vascular inflammation (C-reactive protein), and flow-mediated dilation in the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Medical resident in MICU rotation
* Non-smoker
* Body mass index <28 kg/m2

Exclusion Criteria:

* Systolic blood pressure >140 mmHg; Diastolic blood pressure >90 mmHg
* Known history of diabetes mellitus, hypertension, hyperlipidemia
* Known history of acute or chronic inflammatory or infectious disease
* Known history of sleep disturbance unrelated to work
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2004-12; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Katz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States